CLINICAL TRIAL: NCT03446911
Title: Combining SBRT and Immunotherapy in Early Stage NSCLC Patients Planned for Surgery: Exploring Safety and Immunological Proof of Principle.
Brief Title: Combining SBRT and Immunotherapy in Early Stage NSCLC Patients Planned for Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, A.J. de Langen, Dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MK3475-586
Record Dates: First submitted 2017-11-08; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: NSCLC, Stage I
Keywords: SABR; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SABR (Active Comparator): Patients receive prior to surgery (lobectomy) SABR.
  Interventions: Radiation: SABR
- SABR + pembrolizumab (Active Comparator): Patients receive prior to surgery (lobectomy) SABR + 2 rounds of pembrolizumab
  Interventions: Combination Product: SABR + pembrolizumab

INTERVENTIONS:
Radiation: SABR — Prior to surgery (lobectomy), patients receive stereotactic ablative radiotherapy.
  Arms: SABR
Combination Product: SABR + pembrolizumab — Prior to surgery (lobectomy), patients receive stereotactic ablative radiotherapy + 2 rounds of pembrolizumab
  Arms: SABR + pembrolizumab

SUMMARY:
This study aims to evaluate the safety and mechanisms of action of the trimodality treatment (radiotherapy, immunotherapy and surgery) in early-stage non-small cell lung cancer. Half of the patients will receive stereotactic ablative radiotherapy followed by 2 cycles of immunotherapy (pembrolizumab); the other half will not receive the immunotherapy treatment. After treatment, both groups will continue treatment according to guidelines and will undergo surgery (lobectomy).

DETAILED DESCRIPTION:
An open label randomized exploratory study of the safety and mechanisms of action of combined treatment with SBRT and immunotherapy (pembrolizumab, anti-PD1) for early stage NSCLC.

Intervention:

Patients will be randomized between SBRT with or without 2 cycles of pembrolizumab treatment (starting on the first day of radiotherapy). The patients will undergo a lobectomy with hilar and mediastinal lymph node dissection after SBRT +/- pembrolizumab treatment. Translational research to explore the immune mechanism of action will include biological imaging with immuno-PET (positron emission tomography). Expression rates and activation states of immune effector subsets will be assessed in tumor core biopsy specimens, peripheral blood and tumor draining lymph nodes (TDLNs) by means of fine needle aspirates of TDLNs.

Main study parameters/endpoints:

To assess the safety of combined SBRT and pembrolizumab treatment in early stage NSCLC and to identify the immunological mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed diagnosis of early stage (T1bN0 and T2aN0) peripherally located NCSLC, eligible for surgical resection.
2. Be willing and able to provide written informed consent/assent for the trial.
3. Be 18 years of age or over on day of signing informed consent.
4. Have measurable disease based on RECIST 1.1.
5. Must provide tissue from a core or excisional biopsy of the primary tumor lesion.
6. Have a performance status of 0-1 on the ECOG Performance Scale.
7. Demonstrate adequate organ function, all screening labs should be performed within 10 days of treatment initiation.
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* 1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.

  2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.

  3. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.

  4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

  5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.

  6. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.

  7. Has a history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.

  8. Has an active infection requiring systemic therapy. 9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

  10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

  11. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.

  12. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).

  13. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).

  14. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

  15. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events in patients treated by combining SBRT and pembrolizumab | Up to 90 days post-treatment
  Safety of the combination of SBRT and pembrolizumab will be assessed by the percentage of ≥3 pneumonitis. When combined SBRT and pembrolizumab treatment results in NCIC-CTC grade ≥3 pneumonitis in ≤10% of patients, the combination is regarded as safe. Serious adverse events will be recorded to assess both incidence and severity.

SECONDARY OUTCOMES:
PD-1 expression | Up to 90 days post-treatment
  PD-1 expression in tumor tissue, tumordraining lymphnodes and peripheral blood.
PD-L1 expression | Up to 90 days post-treatment
  PD-L1 expression in tumor tissue, tumordraining lymphnodes and peripheral blood.
CD4 expression | Up to 90 days post-treatment
  CD4 expression in tumor tissue, tumordraining lymphnodes and peripheral blood.
CD8 expression | Up to 90 days post-treatment
  CD8 expression in tumor tissue, TDLN's and peripheral blood.
FoxP3 expression | Up to 90 days post-treatment
  FoxP3 expression in tumor tissue, tumordraining lymphnodes and peripheral blood.
Ki67 expression | Up to 90 days post-treatment
  Ki67 expression in tumor tissue, tumordraining lymphnodes and peripheral blood.
Immune cell count | Up to 90 days post-treatment
  Cell count of the individual immune cells in tumordraining lymphnodes and non-tumordraining lymphnodes
Analysis of PET data - SUVmax (standardized uptake value) | Up to 90 days post-treatment
  SUVmax will be measured in all tumor lesions, enlarged lymph nodes and liver, kidneys, lungs, spleen and left ventricle of the heart.
Analysis of PET data - SUVpeak (standardized uptake value) | Up to 90 days post-treatment
  SUVpeak will be measured in all tumor lesions, enlarged lymph nodes and liver, kidneys, lungs, spleen and left ventricle of the heart.
Analysis of PET data -SUVmean (standardized uptake value) | Up to 90 days post-treatment
  SUVmean will be measured in all tumor lesions, enlarged lymph nodes and liver, kidneys, lungs, spleen and left ventricle of the heart.
Analysis of CT data - Hounsfield Unit density | Up to 90 days post-treatment
  The pre- and post SBRT +/- pembrolizumab CT scans will be assessed for HU density and f-air values
Analysis of CT data - f-air values | Up to 90 days post-treatment
  The pre- and post SBRT +/- pembrolizumab CT scans will be assessed for and f-air values
Correlation between PET data and Blood + Tissue markers | Up to 90 days post-treatment
  The data of the PET-scan will be analyzed and compared to the blood and tissue samples to find a correlation between findings.
Correlation between tumor uptake of Zr89-pembrolizumab and irAEs | Up to 90 days post-treatment
  SUV are values used to describe PET-data. irAE's are specific adverse events. This outcome aims to correlate the (possible) irAE's with the PET-data.

CONTACTS AND LOCATIONS:
Overall Officials: E.F. Smit, MD, PhD, Principal Investigator — The Netherlands Cancer Institute; A.J. de Langen, MD, PhD, Study Chair — The Netherlands Cancer Institute

REFERENCES:
- [Derived] Borm FJ, Smit J, Bakker J, Wondergem M, Smit EF, de Langen AJ, de Gruijl TD. Early response evaluation of PD-1 blockade in NSCLC patients through FDG-PET-CT and T cell profiling of tumor-draining lymph nodes. Oncoimmunology. 2023 Apr 26;12(1):2204745. doi: 10.1080/2162402X.2023.2204745. eCollection 2023. PMID 37123045

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT03446911/Prot_SAP_000.pdf